CLINICAL TRIAL: NCT04773886
Title: To Evaluate the Effectiveness of Mineral Trioxide Aggregate and Platelet Rich Fibrin Along With Biodentine as Pulpotomy Medicament in Patients With Pulpitis.
Brief Title: Effectiveness of Mineral Trioxide Aggregate and Platelet Rich Fibrin Along With Biodentine. .
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, DR SURINDER SACHDEVA, PROFESSOR, Maharishi Markendeswar University (Deemed to be University)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MahrishiMU 1012
Record Dates: First submitted 2021-02-22; First posted 2021-02-26 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Pulpitis - Irreversible
Keywords: pulpal regeneration; pulpitis; pulpotomy
MeSH Terms: conditions — Pulpitis | interventions — mineral trioxide aggregate; Pemetrexed; tricalcium silicate

STUDY DESIGN:
Intervention Model Description: Sixty systemically healthy patients with irreversible pulpitis were enrolled in the study based on inclusion and exclusion criteria. All the enrolled patients were randomly allocated into 4 groups (15 each)
  Group I: MTA GROUP: Vital Pulpotomy will be done using Mineral trioxide aggregate (MTA) as pulp capping agent. Group II: BIODENTINE GROUP: Vital Pulpotomy will be done using Biodentine as pulp capping agent. Group III: PRF + MTA GROUP: Vital Pulpotomy will be done using PRF and Mineral trioxide aggregate (MTA) as pulp capping agent. Group IV: PRF+ BIODENTINE GROUP: Vital Pulpotomy will be done using PRF and Biodentine as pulp capping agent.
Who Masked: Participant, Outcomes Assessor
Masking Description: patient and statistician are masked about the treatment modality.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- MTA GROUP (Sham Comparator): Vital Pulpotomy will be done using Mineral trioxide aggregate(MTA) as pulp capping agent.
  Interventions: Drug: Mineral trioxide aggregate
- BIODENTINE GROUP (Sham Comparator): Vital Pulpotomy will be done using Biodentine as pulp capping agent.
  Interventions: Drug: Biodentine
- PRF + MTA GROUP (Active Comparator): Vital Pulpotomy will be done using PRF and Mineral trioxide aggregate (MTA) as pulp capping agent
  Interventions: Drug: Mineral trioxide aggregate; Biological: Platelet rich fibrin
- PRF+ BIODENTINE GROUP (Active Comparator): Vital Pulpotomy will be done using PRF and Biodentine as pulp capping agent.
  Interventions: Drug: Biodentine; Biological: Platelet rich fibrin

INTERVENTIONS:
Drug: Mineral trioxide aggregate — Vital Pulpotomy will be done using Mineral trioxide aggregate (MTA) as pulp capping agent
  Other Names: MTA
  Arms: MTA GROUP; PRF + MTA GROUP
Drug: Biodentine — Vital Pulpotomy will be done using Biodentine as pulp capping agent
  Other Names: Biodenine
  Arms: BIODENTINE GROUP; PRF+ BIODENTINE GROUP
Biological: Platelet rich fibrin — 10 ml of blood was drawn from the peripheral vein in the selected patients with the help of sterilized disposable syringe and blood was collected in the pre-sterilized borosilicate glass test tube, without any addition of anticoagulant and was immediately centrifuged at 3000 rpm for 15 minutes in a centrifuge unit.
  The product obtained after centrifugation consisted of three layers:
  * Acellular platelet plasma- top most layer
  * Platelet rich fibrin -middle layer
  * Red blood corpuscles- bottom layer PRF was then separated from the red blood corpuscles base with the help of sterile tweezers and scissors and squeezed with the help of sterile gauze piece
  Arms: PRF + MTA GROUP; PRF+ BIODENTINE GROUP

SUMMARY:
The aim of this study was to clinically and radiographically evaluate the effectiveness of MTA, Biodentine, Platelet Rich Fibrin along with Mineral Trioxide Aggregate and Platelet Rich Fibrin along with Biodentine as pulpotomy medicament in patients with pulpitis.

DETAILED DESCRIPTION:
Sixty systemically healthy patients with irreversible pulpitis were enrolled in the study based on inclusion and exclusion criteria. All the enrolled patients were randomly allocated into 4 groups (15 each)

Group I: MTA GROUP: Vital Pulpotomy will be done using Mineral trioxide aggregate (MTA) as pulp capping agent. Group II: BIODENTINE GROUP: Vital Pulpotomy will be done using Biodentine as pulp capping agent. Group III: PRF + MTA GROUP: Vital Pulpotomy will be done using PRF and Mineral trioxide aggregate (MTA) as pulp capping agent. Group IV: PRF+ BIODENTINE GROUP: Vital Pulpotomy will be done using PRF and Biodentine as pulp capping agent Patients were assessed at 1 day,3 months, 6 months and 9 months postoperatively for pain, pulp sensitivity test, swelling or presence of any sinus tract. All the proposed teeth were assessed radiographically at1 day, 3 months, 6 months and 9 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients with carious exposed tooth exhibiting clinical and radiographical evidence for pulpitis.
* Deep caries extending ≥2/3 of dentin.
* Tooth with positive response with cold testing.
* Tooth with no mobility.
* No signs of pulpal necrosis including sinus tract or swelling.
* Patient approval for the treatment and follow up

Exclusion Criteria:

* Any systemic disease that could influence the outcome.
* Non-restorable tooth.
* Teeth with periapical widening.
* Tooth which cannot be isolated.
* Teeth with marginal periodontitis or crestal bone loss.
* Indication of post/ post and core restoration marginal periodontitis with attachment loss >5mm.
* Teeth with immature root or calcified canal.
* Teeth with internal and external resorption.
* No pulp exposure after caries excavation.
* Uncontrolled bleeding after access cavity preparation after several minutes N
* No bleeding at all at the time of access opening
* Pregnant or nursing women.
* Individual hypersensitive or allergic to any product used in the study

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
EPT | change from baseline to 1day, 3 months, 6 months, 9 months
  Electric pulp testing
cold test | change from baseline to 1day, 3 months, 6 months, 9 months
  cold test

SECONDARY OUTCOMES:
Tender on percussion | change from baseline to 1day, 3 months, 6 months, 9 months
  present or absent
swelling | change from baseline to 1day, 3 months, 6 months, 9 months
  present or absent

CONTACTS AND LOCATIONS:
Overall Officials: surinder sachdeva, M.D.S., Study Director — PROFESSOR
Locations (1):
- Department of Conservative Dentistry and Endodontics, M.M. College of Dental Sciences and Research., Ambāla, Haryana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li Y, Sui B, Dahl C, Bergeron B, Shipman P, Niu L, Chen J, Tay FR. Pulpotomy for carious pulp exposures in permanent teeth: A systematic review and meta-analysis. J Dent. 2019 May;84:1-8. doi: 10.1016/j.jdent.2019.03.010. Epub 2019 Apr 11. PMID 30981748
- [Background] Kumar V, Juneja R, Duhan J, Sangwan P, Tewari S. Comparative evaluation of platelet-rich fibrin, mineral trioxide aggregate, and calcium hydroxide as pulpotomy agents in permanent molars with irreversible pulpitis: A randomized controlled trial. Contemp Clin Dent. 2016 Oct-Dec;7(4):512-518. doi: 10.4103/0976-237X.194107. PMID 27994420